CLINICAL TRIAL: NCT06141850
Title: Project PEACH2: Promoting Engagement and COVID-19 Testing for Health
Brief Title: Promoting Engagement and COVID-19 Testing for Health
Acronym: PEACH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Morehouse School of Medicine (Other); Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, Mary Beth Weber, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00006531; 1U01DK132737 (NIH)
Record Dates: First submitted 2023-11-17; First posted 2023-11-21 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project PEACH2 Intervention (Experimental): In addition to a text-based reporting tool for reporting COVID-19 testing, participants randomized to the Project PEACH2 intervention will be sent weekly behavioral nudges via mobile phone text message to encourage adherence to COVID-19 testing and preventive behaviors.
  Interventions: Behavioral: COVID-19 Test Reporting; Behavioral: Personalized Nudges via Text Messaging
- Control Group (Active Comparator): Participants randomized to the control group will receive access to the text-based COVID-19 reporting tool and receive weekly texts on diabetes prevention, management or care.
  Interventions: Behavioral: COVID-19 Test Reporting; Behavioral: Non-personalized Nudges via Text Messaging

INTERVENTIONS:
Behavioral: COVID-19 Test Reporting — Participants will use a simple text-based data reporting tool which they will be asked to use to report any COVID-19 testing during the 12-month long tudy.
Behavioral: Personalized Nudges via Text Messaging — Weekly behavioral nudges via mobile phone text messages, personalized to participants' diabetes status, race/ethnicity, age group, sex, and/or vaccine/testing history, will be sent in weeks 1-16 of the intervention to encourage adherence to COVID-19 testing and preventive behaviors as well as other behaviors important for diabetes management, prevention, or care.
  Arms: Project PEACH2 Intervention
Behavioral: Non-personalized Nudges via Text Messaging — Weekly behavioral nudges via mobile phone text messages will be sent in weeks 1-16 of the intervention sharing tips lifestyle behaviors important for diabetes management and prevention (e.g., exercise, eating a healthy diet, etc.).
  Arms: Control Group

SUMMARY:
PEACH2 is a community-based study, targeting individuals affected by diabetes. Study participants will be randomized into the PEACH2 Intervention Arm or the Control Arm. The intervention lasts for 16 weeks and participants will be followed for 12 months in total.

DETAILED DESCRIPTION:
This study leverages data collected during Project PEACH 1: Promoting Engagement and COVID-19 Testing for Health, a Rapid Acceleration of Diagnostics - Underserved Populations (RADx-UP) funded study to understand barriers to effective and equitable coronavirus disease 2019 (COVID-19) testing in high-risk and minority populations in Georgia that are affected by diabetes. PEACH 1 applied mixed-methods (quantitative, qualitative, geographic and spatial analysis) to gather evidence to describe COVID-19 epidemiology, locate regions and populations with low testing and vaccine uptake, and targeting key informant interviewing and monitoring social and news media, to identify barriers, motivators, and perceptions around COVID-19 as well as related behaviors among different populations and regions.

Analysis of Project PEACH 1 data collected from key informants and community partners indicated gaps in capacity for and commitment to community testing when vaccines became available, and sites were pivoting to prioritize vaccinations even as they continued to provide COVID-19 testing. However, COVID-19 testing can be a key tool to address the pandemic, particularly in areas with low vaccination rates and high diabetes rates such as Georgia. People with diabetes, prediabetes, and obesity have elevated risk for COVID-19 infection and are more likely to suffer in-hospital complications. Further, Diabetes is 2.4 times more common in socioeconomically vulnerable and minority populations. Throughout the pandemic, counties with predominantly Black communities had a 6-fold COVID-19 death rate compared to those that are predominantly White. For these reasons, finding sustainable, easy to disseminate, and acceptable ways to increase and sustain COVID-19 testing is needed. Further, understanding the relationship between attitudes toward testing in situations of continued vaccine hesitancy and resistance and developing insights in how to address them in a dynamic pandemic situation will be fundamental to future pandemic response.

COVID-19 testing, both home-based testing and clinic testing, must remain a key feature for diabetes management and prevention to reduce secondary complications associated with infection. Home-based testing may help people overcome barriers to testing (identifying where to get tested, scheduling and attending appointments, stigma). However, in order for it to be successful there is a need to understand the feasibility, acceptability, and sustainability of at-home testing as well as the perceived advantages and disadvantages of home-based testing compared to clinic-based testing among the high-risk population of individuals affected by or at risk for diabetes. This information can be used to create targeted behavioral "nudges". Nudges are indirect suggestions and positive reinforcements designed to encourage certain choices. They may be a useful means of promoting acceptability and usage of COVID-19 testing as well as increasing an understanding of and acceptability of other key preventive behaviors like COVID-19 vaccination. Behavioral nudges have been shown to have a noticeable effect on health behaviors and study recruitment, however, research testing the application of behavioral nudges relating to behavior change around disease prevention in a pandemic situation is needed.

Study participants will be randomized into the PEACH2 Intervention Arm or the Control Arm. At baseline, all participants will be asked to complete a baseline survey to collect demographic data, history of COVID-19, diabetes, and diabetes risk factors, views of COVID-19, COVID-19 preventive behaviors (including vaccination), and experiences with COVID-19 testing. Participants will be asked to report, using a simple text-based data reporting tool, any COVID-19 testing during the 12-month study. Participants are administered surveys at Baseline, after completing the 16 week intervention and at Month 12 to collect information on COVID-19 testing, prevention, and vaccine behaviors and views.

In addition, Project PEACH2 Intervention participants will be sent weekly personalized behavioral nudges via mobile phone text message during the 16 week long intervention to encourage adherence to COVID-19 testing and preventive behaviors as well as share important tips for diabetes management, prevention or care. Nudges targeting testing behaviors will be delivered whereby participants who have not reported (1) having symptoms indicative of a possible infection with a viral disease and (2) a COVID-19 test in the past four weeks will receive a nudge to encourage COVID-19 testing. Other behavioral nudges will target other COVID-19 related preventive behaviors (e.g., staying home when sick, wear a mask, etc.) and diabetes management/prevention/care behaviors (e.g., increasing physical activity, improving diet, decreasing stress, etc). Nudge personalization targeting relationship with diabetes, age group, sex, vaccine and testing history, and race/ethnicity will be based on data collected in PEACH 1 as well as ongoing social media and data analysis in PEACH2.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Living in Georgia, USA
* Have access to a cellphone
* Not currently pregnant
* At-risk for diabetes, have diabetes, or are a family caregiver of someone living with diabetes
* Agree to receive text messages and be randomized to the intervention or control arm of the study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Percent of Participants Using a COVID-19 Test | Baseline, Weeks 4, 8, 12, and 16
  The percent of individuals reporting taking a COVID-19 test in the past month as reported using the text-based COVID-19 reporting tool created for this study.

SECONDARY OUTCOMES:
Frequency of Taking a COVID-19 Test | Baseline, Weeks 4, 8, 12, and 16
  The frequency of COVID-19 testing as reported using the text-based COVID-19 reporting tool created for this study.
Number of Participants Receiving Annual COVID-19 Vaccination | Baseline, Week 16 (completion of intervention), and Month 12
  The number of participants receiving a partial or full dose of an approved COVID-19 vaccination.
Number of Participants Adhering to COVID-19 Prevention Behaviors | Baseline, Week 16 (completion of intervention), and Month 12
  The number of participants reporting adhering to COVID-19 prevention behaviors is assessed based on survey responses on questions about masking, social distancing, isolating/quarantining when needed, and vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Weber, PhD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All deidentified data will be made publicly available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available upon trial completion, with no end date.
Access Criteria: Data will be available to anyone who wishes to access the data, for any purpose. Data will be available by emailing the study PI at mbweber@emory.edu or though the data repositories for the RADx-UP network.

DOCUMENTS (1):
  • Informed Consent Form (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT06141850/ICF_000.pdf